CLINICAL TRIAL: NCT01268059
Title: A Phase 1b/2 Randomized Study of MEDI-575 in Combination With Carboplatin Plus Paclitaxel Versus Carboplatin Plus Paclitaxel Alone in Adult Subjects With Previously Untreated, Advanced Non-Small Cell Lung Cancer
Brief Title: A Study of Carboplatin and Paclitaxel With or Without MEDI-575 in Untreated, Advanced Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: In conjunction with the overall risk-benefit assessment, study was terminated prematurely due to safety concerns.
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CD-ON-MEDI-575-1031
Record Dates: First submitted 2010-12-17; First posted 2010-12-29 (Estimated); Results first posted 2020-12-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-11

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small cell lung cancer; NSCLC; MEDI-575; Platelet-derived growth factor receptor alpha
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Paclitaxel; Tovetumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carboplatin/Paclitaxel (Active Comparator): Carboplatin/paclitaxel regimen (carboplatin area under the plasma concentration-time curve [AUC] of 6 milligram per milliliter into minute [mg/mL*min], and paclitaxel 200 milligram per square meter [mg/m^2]) administered as an intravenous (IV) infusion once every 21 days on Day 1, for a total of 6 doses (cycles) until unacceptable toxicity, disease progression, or other reasons for participant withdrawal. Subjects were enrolled from North America/European Union (EU) and Japan regions.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel
- Carboplatin/Paclitaxel + MEDI-575 (Experimental): Carboplatin/paclitaxel regimen (carboplatin AUC = 6 mg/mL*min, and paclitaxel 200 mg/m^2) followed by MEDI-575 at a dose of 25 milligram per kilogram (mg/kg) administered as an IV infusion once every 21 days on Day 1 for a total of 6 cycles until unacceptable toxicity, disease progression, initiation of alternative anticancer therapy, or other reasons for participant withdrawal. MEDI-575 alone continued in those participants who achieved stable disease or better at the completion of carboplatin/paclitaxel therapy and did not demonstrate toxicity to MEDI-575. Subjects were enrolled from North America/European Union (EU) and Japan regions.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: MEDI-575

INTERVENTIONS:
Drug: Carboplatin — Carboplatin (carboplatin area under the plasma concentration-time curve [AUC] of 6 milligram per milliliter into minute [mg/mL*min] administered as an intravenous (IV) infusion once every 21 days on Day 1, for a total of 6 doses (cycles) until unacceptable toxicity, disease progression, or other reasons for participant withdrawal.
Drug: Paclitaxel — Paclitaxel 200 milligram per square meter (mg/m^2) administered as an intravenous (IV) infusion once every 21 days on Day 1, for a total of 6 doses (cycles) until unacceptable toxicity, disease progression, or other reasons for participant withdrawal.
Drug: MEDI-575 — MEDI-575 at a dose of 25 milligram per kilogram (mg/kg) administered as an IV infusion once every 21 days on Day 1 for a total of 6 cycles until unacceptable toxicity, disease progression, initiation of alternative anticancer therapy, or other reasons for participant withdrawal. MEDI-575 alone continued in those participants who achieved stable disease or better at the completion of carboplatin/paclitaxel therapy and did not demonstrate toxicity to MEDI-575.
  Arms: Carboplatin/Paclitaxel + MEDI-575

SUMMARY:
The purpose of this study is to evaluate the dose, antitumor activity, safety and pharmacology of MEDI-575 in combination with carboplatin/paclitaxel in subjects with previously untreated, advanced non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
This is a Phase 1b/2, multicenter, open-label study of MEDI-575 to evaluate the dose, anti-tumor activity, safety, and pharmacology (pharmacokinetics, immunogenicity, and biomarkers) of MEDI-575 in combination with carboplatin/paclitaxel in subjects with previously untreated, advanced non-small cell lung cancer. This study has two phases: dose determination (Phase 1b) and randomization (Phase 2).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed inoperable Stage IIIB or Stage IV non-small cell lung cancer according to the Seventh Edition of the American Joint Committee on Cancer (AJCC) Tumor Node Metastases (TNM) staging system (only participants with squamous cell carcinoma will be enrolled)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy of greater than or equal to (>=) 3 months
* Prothrombin time elevation less than or equal to (<=) Grade 2 by National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) criteria (Version 4.0) is acceptable for participants on anticoagulant therapy
* Adequate hematologic function
* Adequate organ function
* Suitable candidates for therapy with carboplatin/paclitaxel
* Participants must have at least 1 lesion that is measurable using Response Evaluation Criteria for Solid Tumors
* Participants must be willing to consent to allow collection of archived NSCLC tumor samples
* Negative serum beta-human chorionic gonadotropin (beta-hCG) test (women of childbearing potential only)
* Females of childbearing potential, unless surgically sterile has a sterile male partner, is premenarchal or at least 2 years postmenopausal, or practices abstinence, must use 2 effective methods of avoiding pregnancy (including oral, transdermal, or implanted contraceptives, intrauterine device, female condom with spermicide, diaphragm with spermicide, cervical cap, or use of a condom with spermicide by the sexual partner) from screening, and must agree to continue using such precautions for 90 days after the final dose of treatment; cessation of birth control after this point should be discussed with a responsible physician
* Males, unless surgically sterile, must use 2 effective methods of birth control with a female partner and must agree to continue using such contraceptive precautions from screening through 90 days after the final dose of treatment

Exclusion Criteria:

* At discretion of the investigator regarding safety of the participants
* Concurrent enrollment in another clinical study
* Any concurrent chemotherapy, radiotherapy, immunotherapy, biologic, or hormonal therapy for treatment of cancer
* Previous monoclonal antibody (mAb) treatment specifically directed against platelet-derived growth factor (PDGF) or PDGF receptors
* History of serious allergy or reaction to any component of the MEDI-575 formulation
* Receipt of any previous systemic anticancer therapies for advanced or metastatic disease
* Previous adjuvant/neoadjuvant radiotherapy or chemotherapy for treatment of previous nonmetastatic disease is allowed provided that 6 months have elapsed from the end of such therapies to the time of enrollment
* New York Heart Association >= Class II congestive heart failure
* History of myocardial infarction, unstable angina, transient ischemic attack or stroke within the previous 6 months prior to enrollment
* History of other invasive malignancy within 5 years except for cervical carcinoma in situ (CIS), non-melanomatous carcinoma of the skin or ductal carcinoma in situ (DCIS) of the breast that have been surgically cured
* Evidence of active infection requiring the use of systemic antimicrobial treatment within 72 hours prior to initial treatment with MEDI-575
* Use of immunosuppressive medication (inhaled and topical corticosteroids are permitted) within 7 days prior to enrollment
* Systemic immunosuppressive steroid therapy
* Participants may take replacement doses of steroids if on a stable dose for at least 2 weeks prior to enrollment
* History of active human immunodeficiency virus (HIV) or active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
* Pregnancy or lactation
* Previous medical history or evidence of an inter-current illness
* Any physical, social, or psychiatric condition which would prevent effective cooperation or participation in the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2010-12-16 (Actual); Primary Completion 2013-09-11 (Actual); Study Completion 2013-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MedImmune LLC, Study Director — MedImmune LLC
Locations (28):
- United States (18):
  - Research Site, Fountain Valley, California
  - Research Site, Oxnard, California
  - Research Site, Chicago, Illinois
  - Research Site, Lafayette, Indiana
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Annapolis, Maryland
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Danvers, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Omaha, Nebraska
  - Research Site, Lake Success, New York
  - Research Site, Canton, Ohio
  - Research Site, Hershey, Pennsylvania
  - Research Site, Hilton Head Island, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Corpus Christi, Texas
  - Research Site, Houston, Texas
- Research Site, Ottawa, Ontario, Canada
- Research Site, Marseille, France
- Research Site, Berlin, Germany
- Research Site, Szombathely, Hungary
- Japan (2):
  - Research Site, Fukuoka
  - Research Site, Sunto-gun
- Poland (4):
  - Research Site, Gdansk
  - Research Site, Lodz
  - Research Site, Mrozy
  - Research Site, Szczecin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Overall, 99 participants were enrolled in the study, (4 participants, all from North America sites, were enrolled in the Phase 1b part of the study and 95 participants in Phase 2 part of the study). Of 95 participants, 14 were enrolled from Japan sites, and 81 were from North American and European Union (EU) sites.
Groups:
- Carboplatin/Paclitaxel (C/P): North America/EU Population: Carboplatin/paclitaxel regimen (carboplatin area under the plasma concentration-time curve [AUC] of 6 milligram per milliliter into minute [mg/mL*min], and paclitaxel 200 milligram per square meter [mg/m^2]) administered as an intravenous (IV) infusion once every 21 days on Day 1, for a total of 6 doses (cycles) or until unacceptable toxicity, disease progression, or other reasons for participant withdrawal.
- C/P + MEDI-575 (C/P/M): North America/EU Population; C/P + MEDI-575 (C/P/M): Japan Population: Carboplatin/paclitaxel regimen (carboplatin AUC = 6 mg/mL*min, and paclitaxel 200 mg/m^2) followed by MEDI-575 at a dose of 25 milligram per kilogram (mg/kg) administered as an IV infusion once every 21 days on Day 1 for a total of 6 cycles. Participants who achieved stable disease or better at the completion of carboplatin/paclitaxel therapy and did not demonstrate toxicity to MEDI-575, MEDI-575 alone was continued until unacceptable toxicity, disease progression, initiation of alternative anticancer therapy, or other reasons for participant withdrawal.
- Carboplatin/Paclitaxel (C/P): Japan Population: Carboplatin/paclitaxel regimen (carboplatin AUC = 6 mg/mL*min, and paclitaxel 200 mg/m^2) administered as an IV infusion once every 21 days on Day 1, for a total of 6 doses (cycles) or until unacceptable toxicity, disease progression, or other reasons for participant withdrawal.
Period: Overall Study
Arm/Group | Carboplatin/Paclitaxel (C/P): North America/EU Population | C/P + MEDI-575 (C/P/M): North America/EU Population | Carboplatin/Paclitaxel (C/P): Japan Population | C/P + MEDI-575 (C/P/M): Japan Population
Started | 40 | 45 (Arm applicable for both dose-determination (Phase 1b) and randomization phase (Phase 2) of study.) | 6 | 8
Completed | 12 (End of study defined as 14 months from the last participant enrolled, or sponsor stopped the study.) | 10 (End of study defined as 14 months from the last participant enrolled, or sponsor stopped the study.) | 3 (End of study defined as 14 months from the last participant enrolled, or sponsor stopped the study.) | 3 (End of study defined as 14 months from the last participant enrolled, or sponsor stopped the study.)
Not Completed | 28 | 35 | 3 | 5
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 4 | 0 | 0
Not completed — Death | 20 | 30 | 3 | 5
Not completed — Progression of disease | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) North America/European Union (EU) population included all North America/EU participants who entered into Phase 1b or were randomized into Phase 2 portion of the study. The ITT Japanese population included all Japanese participants who were randomized into the Phase 2 portion of the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Carboplatin/Paclitaxel (C/P): North America/EU Population | C/P + MEDI-575 (C/P/M): North America/EU Population | Carboplatin/Paclitaxel (C/P): Japan Population | C/P + MEDI-575 (C/P/M): Japan Population | Total
Number analyzed (Participants) | 40 | 45 | 6 | 8 | 99
Age, Customized [Count of Participants; unit: Participants]
  less than or equal to (<=) 70 years | 35 (6.6) | 32 (8.2) | 6 (13.9) | 6 (6.0) | 79
  greater than (>) 70 years | 5 | 13 | 0 | 2 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 2 | 2 | 38
  Male | 23 | 28 | 4 | 6 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 0 | 3
  Not Hispanic or Latino | 39 | 43 | 6 | 8 | 96
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 6 | 8 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 5 | 0 | 0 | 8
  White | 37 | 39 | 0 | 0 | 76
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLT): Phase 1b
Description: A DLT was defined as:
  1. Any treatment-related Grade 3 or higher non-hematologic toxicity that occurred during the DLT assessment period with the following exceptions:
     1. Grade 3 fever (in the absence of neutropenia) defined as more than (>) 40.0 degree Celcius (> 104.0 degree Fahrenheit) that resolved to normal or baseline within 24 hours of treatment and was not considered a serious adverse event (SAE); or
     2. Grade 3 rigors/chills that responded to optimal therapy.
  2. Any treatment-related Grade 3 or higher hematologic toxicity.
Time Frame: From Day 1 to Day 21 of first cycle
Population: The evaluable population for dose determination included all participants who were in Phase 1b, received at least 1 full cycle of MEDI-575 and completed the safety follow-up through the DLT evaluation period or participants who experienced any DLT.
Measure: Count of Participants; unit: Participants
Groups:
- Carboplatin/Paclitaxel + MEDI-575 - Phase 1b: Carboplatin/paclitaxel regimen (carboplatin AUC = 6 mg/mL*min, and paclitaxel 200 mg/m^2) followed by MEDI-575 at a dose of 25 milligram per kilogram (mg/kg) administered as an IV infusion once every 21 days on Day 1 for a total of 6 cycles. Participants who achieved stable disease or better at the completion of carboplatin/paclitaxel therapy and did not demonstrate toxicity to MEDI-575, MEDI-575 alone was continued until unacceptable toxicity, disease progression, initiation of alternative anticancer therapy, or other reasons for participant withdrawal.
Arm/Group | Carboplatin/Paclitaxel + MEDI-575 - Phase 1b
Number analyzed (Participants) | 4
Participants | 0

2. Primary Outcome: Progression Free-Survival (PFS)
Description: Progression-free survival defined as the time from randomization (randomization referred to the date of treatment assignment) to disease progression (defined according to Response Evaluation Criteria for Solid Tumors [RECIST] version 1.1 guidelines) or death due to any cause, whichever occurs first. Participants without progression or death at the time of analysis were censored at their last date of tumor evaluation. PFS was assessed only in North America/European Union (EU) participants. Progression-free survival was evaluated using Kaplan-Meier method.
Time Frame: From randomization until the end of study (14 months from last participant enrolled or sponsor stopped the study), assessed at every 6 weeks until disease progression and every 3 months until the end of the study (approximately 3 years)
Population: The Intent-to-Treat (ITT) North America/EU population included all North America/EU participants who were randomized into Phase 2 portion of the study. The PFS was analyzed for only those participants who had disease progression.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Carboplatin/Paclitaxel - North America/European Union (EU): Carboplatin/paclitaxel regimen (carboplatin area under the plasma concentration-time curve [AUC] of 6 milligram per milliliter into minute [mg/mL*min], and paclitaxel 200 milligram per square meter [mg/m^2]) administered as an intravenous (IV) infusion once every 21 days on Day 1, for a total of 6 doses (cycles) or until unacceptable toxicity, disease progression, or other reasons for participant withdrawal.
- Carboplatin/Paclitaxel + MEDI-575 - North America/EU: Carboplatin/paclitaxel regimen (carboplatin AUC = 6 mg/mL*min, and paclitaxel 200 mg/m^2) followed by MEDI-575 at a dose of 25 milligram per kilogram (mg/kg) administered as an IV infusion once every 21 days on Day 1 for a total of 6 cycles. Participants who achieved stable disease or better at the completion of carboplatin/paclitaxel therapy and did not demonstrate toxicity to MEDI-575, MEDI-575 alone was continued until unacceptable toxicity, disease progression, initiation of alternative anticancer therapy, or other reasons for participant withdrawal.
Arm/Group | Carboplatin/Paclitaxel - North America/European Union (EU) | Carboplatin/Paclitaxel + MEDI-575 - North America/EU
Number analyzed (Participants) | 19 | 27
months | 5.5 [4.7 to 6.5] | 4.6 [3.9 to 5.5]
Statistical Analysis 1: Comparison: Carboplatin/Paclitaxel - North America/European Union (EU) vs Carboplatin/Paclitaxel + MEDI-575 - North America/EU; Test type: Superiority or Other; p = 0.027, Log Rank; The 2-sided p-value was calculated using the log-rank test stratified by histology, disease stage, and ECOG performance status; Hazard Ratio (HR) = 2.205, 95% CI 2-sided [1.1 to 4.5] — Hazard ratio and its 95 percent (%) confidence interval ( CIs) were calculated using the Cox proportional hazard model stratified by histology, disease stage, and Eastern Cooperative Oncology Group (ECOG) performance status

3. Secondary Outcome: Best Overall Response
Description: Best overall response of a participant was defined as the best tumor response [Complete Response (CR), Partial Response (PR), Stable Disease (SD), or Progressive Disease (PD)] observed during the trial period assessed according to the Response Evaluation Criteria for Solid Tumors (RECIST) version 1.1 criteria. The participant's best overall response assignment depended on the findings of both target and non-target disease and also on the appearance of new lesions. CR was defined as disappearance of tumor lesions, PR was defined as a decrease of at least 30 percent (%) in the sum of diameters of target lesion, SD was defined as steady state of disease, and PD was defined as an increase of at least 20% in the sum of diameters of target lesions.
Time Frame: From initiation of treatment until the end of study (14 months from last participant enrolled or sponsor stopped the study), assessed at every 6 weeks until disease progression and every 3 months until the end of the study (approximately 3 years)
Population: The ITT North America/European Union (EU) population included all North America/EU participants who were randomized into Phase 2 portion of the study. The ITT Japanese population included all Japanese participants who were randomized into the Phase 2 portion of the study.
Measure: Count of Participants; unit: Participants
Groups:
- Carboplatin/Paclitaxel - Japan: Carboplatin/paclitaxel regimen (carboplatin area under the plasma concentration-time curve [AUC] of 6 milligram per milliliter into minute [mg/mL*min], and paclitaxel 200 milligram per square meter [mg/m^2]) administered as an intravenous (IV) infusion once every 21 days on Day 1, for a total of 6 doses (cycles) or until unacceptable toxicity, disease progression, or other reasons for participant withdrawal.
- Carboplatin/Paclitaxel + MEDI-575 - Japan: Carboplatin/paclitaxel regimen (carboplatin AUC = 6 mg/mL*min, and paclitaxel 200 mg/m^2) followed by MEDI-575 at a dose of 25 milligram per kilogram (mg/kg) administered as an IV infusion once every 21 days on Day 1 for a total of 6 cycles. Participants who achieved stable disease or better at the completion of carboplatin/paclitaxel therapy and did not demonstrate toxicity to MEDI-575, MEDI-575 alone was continued until unacceptable toxicity, disease progression, initiation of alternative anticancer therapy, or other reasons for participant withdrawal.
Arm/Group | Carboplatin/Paclitaxel - North America/European Union (EU) | Carboplatin/Paclitaxel + MEDI-575 - North America/EU | Carboplatin/Paclitaxel - Japan | Carboplatin/Paclitaxel + MEDI-575 - Japan
Number analyzed (Participants) | 40 | 41 | 6 | 8
Participants
  Complete response | 1 | 0 | 0 | 0
  Partial response | 12 | 19 | 2 | 1
  Stable disease | 19 | 12 | 3 | 5
  Progressive disease | 1 | 5 | 1 | 1
  Unknown | 7 | 5 | 0 | 1

4. Secondary Outcome: Objective Response Rate (ORR)
Description: The ORR defined as the percentage of participants with confirmed CR or confirmed PR according to RECIST version 1.1 guidelines. Confirmed responses were those that persist on repeat imaging or assessment greater than or equal to (>=) 4 weeks after the initial documentation of response. The ORR was evaluated using Kaplan-Meier method.
Time Frame: as for outcome 3
Population: The ITT North America/EU population included all North America/EU participants who were randomized into Phase 2 portion of the study. The ITT Japanese population included all Japanese participants who were randomized into the Phase 2 portion of the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Carboplatin/Paclitaxel - North America/European Union (EU) | Carboplatin/Paclitaxel + MEDI-575 - North America/EU | Carboplatin/Paclitaxel - Japan | Carboplatin/Paclitaxel + MEDI-575 - Japan
Number analyzed (Participants) | 40 | 41 | 6 | 8
percentage of participants | 22.5 [10.8 to 38.5] | 31.7 [18.1 to 48.1] | 33.3 [4.3 to 77.7] | 12.5 [0.3 to 52.7]
Statistical Analysis 1: Comparison: Carboplatin/Paclitaxel - North America/European Union (EU) vs Carboplatin/Paclitaxel + MEDI-575 - North America/EU; Treatment effect Carboplatin/Paclitaxel + MEDI-575 versus Carboplatin/Paclitaxel; Test type: Superiority or Other; p = 0.487, Cochran-Mantel-Haenszel — The 2-sided p-value was calculated by adjusting for the stratification factors histology, disease stage, and Eastern Cooperative Oncology Group (ECOG) performance status
Statistical Analysis 2: Comparison: Carboplatin/Paclitaxel - Japan vs Carboplatin/Paclitaxel + MEDI-575 - Japan; Treatment effect Carboplatin/Paclitaxel + MEDI-575 versus Carboplatin/Paclitaxel; Test type: Superiority or Other; p = 0.386, Cochran-Mantel-Haenszel — The 2-sided p-value was calculated by adjusting for the stratification factors histology, disease stage, and ECOG performance status

5. Secondary Outcome: Time to Response (TTR)
Description: The TTR was measured from initiation of study treatment to the first documentation of objective response (OR). The OR defined as the participants with confirmed CR or confirmed PR according to RECIST version 1.1 guidelines. Confirmed responses were those that persist on repeat imaging or assessment >=4 weeks after the initial documentation of response. The TTR was evaluated using Kaplan-Meier method.
Time Frame: as for outcome 3
Population: The ITT North America/EU population included all North America/EU participants who were randomized into Phase 2 portion of the study. The ITT Japanese population included all Japanese participants who were randomized into the Phase 2 portion of the study. Participants who achieved OR were analyzed for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carboplatin/Paclitaxel - North America/European Union (EU) | Carboplatin/Paclitaxel + MEDI-575 - North America/EU | Carboplatin/Paclitaxel - Japan | Carboplatin/Paclitaxel + MEDI-575 - Japan
Number analyzed (Participants) | 9 | 13 | 2 | 1
months | 1.4 [1.2 to 2.7] | 1.4 [1.3 to 1.6] | 2.2 [1.4 to 3.1] | 2.8 [NA to NA] — The 95% confidence interval was not determined as only 1 participant was analyzed.

6. Secondary Outcome: Duration of Response (DR)
Description: The DR defined as the duration from the first documentation of OR to the first documented disease progression. Participants without progression at the time of analysis were censored at their last date of tumor evaluation. The DR was evaluated using Kaplan-Meier method.
Time Frame: as for outcome 3
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carboplatin/Paclitaxel - North America/European Union (EU) | Carboplatin/Paclitaxel + MEDI-575 - North America/EU | Carboplatin/Paclitaxel - Japan | Carboplatin/Paclitaxel + MEDI-575 - Japan
Number analyzed (Participants) | 9 | 13 | 2 | 1
months | 3.3 [1.3 to 4.6] | 4.2 [3.7 to 5.0] | 4.9 [3.5 to 6.3] | 2.1 [NA to NA] — The 95% confidence interval was not determined as only 1 participant was analyzed.

7. Secondary Outcome: Time to Progression (TTP)
Description: The TTP was measured from randomization until the documentation of disease progression. Disease progression defined according to RECIST version 1.1 guidelines. Participants without progression at the time of analysis were censored at their last date of tumor evaluation. The TTP was evaluated using Kaplan-Meier method.
Time Frame: as for outcome 3
Population: The ITT North America/EU population included all North America/EU participants who were randomized into Phase 2 portion of the study. The ITT Japanese population included all Japanese participants who were randomized into the Phase 2 portion of the study. The TTP was analyzed for only those participants who had disease progression.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carboplatin/Paclitaxel - North America/European Union (EU) | Carboplatin/Paclitaxel + MEDI-575 - North America/EU | Carboplatin/Paclitaxel - Japan | Carboplatin/Paclitaxel + MEDI-575 - Japan
Number analyzed (Participants) | 13 | 23 | 5 | 6
months | 6.4 [4.9 to 10.3] | 4.6 [3.9 to 6.4] | 6.5 [1.4 to 10.7] | 4.6 [1.3 to 15.0]
Statistical Analysis 1: Comparison: Carboplatin/Paclitaxel - North America/European Union (EU) vs Carboplatin/Paclitaxel + MEDI-575 - North America/EU; Test type: Superiority or Other; Hazard Ratio (HR) = 3.017, 95% CI 2-sided [1.2 to 7.4] — The 95% confidence interval calculated using the Cox proportional hazard model stratified by histology, disease stage, and ECOG performance status
Statistical Analysis 2: Comparison: Carboplatin/Paclitaxel - Japan vs Carboplatin/Paclitaxel + MEDI-575 - Japan; Test type: Superiority or Other; Hazard Ratio (HR) = 1.134, 95% CI 2-sided [0.3 to 4.3] — [estimate comment as in outcome 7, analysis 1]

8. Secondary Outcome: Overall Survival (OS)
Description: Overall survival defined as the time from initiation of study treatment until death due to any cause. Participants who were still alive at the time of analysis were censored at their last date of last contact. The OS was evaluated using Kaplan-Meier method.
Time Frame: as for outcome 3
Population: The ITT North America/EU population and the ITT Japanese population included all participants who were randomized into the Phase 2 portion of the study. The "Number of Participants Analyzed" denotes the number of participants evaluated for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carboplatin/Paclitaxel - North America/European Union (EU) | Carboplatin/Paclitaxel + MEDI-575 - North America/EU | Carboplatin/Paclitaxel - Japan | Carboplatin/Paclitaxel + MEDI-575 - Japan
Number analyzed (Participants) | 20 | 27 | 3 | 5
months | 11.8 [8.2 to NA] — Upper 95% CI data not determined as an insufficient number of participants had the event. | 10.0 [6.4 to 11.6] | NA [4.3 to NA] — Median and upper 95% CI data not determined as an insufficient number of participants had the event. | 11.5 [2.3 to NA] — Upper 95% CI data not determined as an insufficient number of participants had the event.
Statistical Analysis 1: Comparison: Carboplatin/Paclitaxel - North America/European Union (EU) vs Carboplatin/Paclitaxel + MEDI-575 - North America/EU; Test type: Superiority or Other; Hazard Ratio (HR) = 1.315, 95% CI 2-sided [0.7 to 2.4] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Carboplatin/Paclitaxel - Japan vs Carboplatin/Paclitaxel + MEDI-575 - Japan; Test type: Superiority or Other; Hazard Ratio (HR) = 2.083, 95% CI 2-sided [0.4 to 10.8] — [estimate comment as in outcome 7, analysis 1]

9. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: From signing of informed consent form until 90 days post the last dose treatment (approximately 3 years)
Population: The safety population included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Carboplatin/Paclitaxel (Total): Carboplatin/paclitaxel regimen (carboplatin area under the plasma concentration-time curve [AUC] of 6 milligram per milliliter into minute [mg/mL*min], and paclitaxel 200 milligram per square meter [mg/m^2]) administered as an intravenous (IV) infusion once every 21 days on Day 1, for a total of 6 doses (cycles) or until unacceptable toxicity, disease progression, or other reasons for participant withdrawal.
- Carboplatin/Paclitaxel + MEDI-575 (Total): Carboplatin/paclitaxel regimen (carboplatin AUC = 6 mg/mL*min, and paclitaxel 200 mg/m^2) followed by MEDI-575 at a dose of 25 milligram per kilogram (mg/kg) administered as an IV infusion once every 21 days on Day 1 for a total of 6 cycles. Participants who achieved stable disease or better at the completion of carboplatin/paclitaxel therapy and did not demonstrate toxicity to MEDI-575, MEDI-575 alone was continued until unacceptable toxicity, disease progression, initiation of alternative anticancer therapy, or other reasons for participant withdrawal.
Arm/Group | Carboplatin/Paclitaxel (Total) | Carboplatin/Paclitaxel + MEDI-575 (Total)
Number analyzed (Participants) | 43 | 53
Participants
  Any AE | 42 | 53
  Any SAE | 17 | 25

10. Secondary Outcome: Number of Participants With Abnormalities in Laboratory Investigations Reported as AEs or SAEs
Description: Laboratory investigations included hematology, coagulation, serum chemistry and urinalysis parameters. Participants with abnormalities in these laboratory investigations recorded as AEs or SAEs were reported.
Time Frame: From signing of informed consent form until 90 days post the last dose treatment (approximately 3 years)
Population: The safety population included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Carboplatin/Paclitaxel (Total) | Carboplatin/Paclitaxel + MEDI-575 (Total)
Number analyzed (Participants) | 43 | 53
Participants
  Anaemia | 15 | 25
  Febrile neutropenia | 3 | 6
  Idiopathic thrombocytopenic purpura | 0 | 1
  Leukopenia | 2 | 6
  Lymphadenopathy | 0 | 2
  Lymphopenia | 2 | 1
  Neutropenia | 7 | 13
  Thrombocytopenia | 3 | 10
  Activated partial thromboplastin time prolonged | 0 | 1
  Haemoglobin decreased | 1 | 5
  Lymphocyte count decreased | 0 | 1
  Neutrophil count decreased | 5 | 14
  Platelet count decreased | 5 | 9
  White blood cell count decreased | 4 | 10
  Alanine aminotransferase increased | 2 | 5
  Aspartate aminotransferase increased | 3 | 4
  Blood alkaline phosphatase increased | 2 | 2
  Blood bilirubin increased | 2 | 0
  Blood creatinine increased | 1 | 3
  Blood magnesium decreased | 0 | 1
  Gamma-glutamyl transferase increased | 0 | 1
  Electrolyte imbalance | 1 | 0
  Hypercholesterolaemia | 1 | 0
  Hyperglycaemia | 5 | 7
  Hypertriglyceridaemia | 2 | 1
  Hypoalbuminaemia | 3 | 7
  Hypocalcaemia | 3 | 6
  Hypoglycaemia | 1 | 1
  Hypokalemia | 8 | 12
  Hypomagnesaemia | 10 | 20
  Hyponatraemia | 4 | 8
  Hypophosphataemia | 2 | 4
  Iron deficiency | 0 | 1
  Vitamin B12 deficiency | 0 | 1
  Urine analysis abnormal | 0 | 1
  Specific gravity urine increased | 0 | 1
  Haematuria | 1 | 1
  Proteinuria | 1 | 1
  Pyelocaliectasis | 0 | 1

11. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities Reported as AEs
Description: The 12-lead ECG data were performed and obtained in triplicate that is 3 ECGs obtained within a 5 minute time period. Number of participants with ECG abnormalities were reported and recorded as AEs.
Time Frame: From signing of informed consent form until 90 days post the last dose treatment (approximately 3 years)
Population: The safety population included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Carboplatin/Paclitaxel (Total) | Carboplatin/Paclitaxel + MEDI-575 (Total)
Number analyzed (Participants) | 43 | 53
Participants
  Atrial fibrillation | 0 | 1
  Atrial flutter | 0 | 1
  Atrioventricular block first degree | 0 | 1
  Myocardial infarction | 1 | 0
  Tachycardia | 2 | 3

12. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of MEDI-575 After First Dose
Description: The Cmax of MEDI-575 after first dose is reported.
Time Frame: Day 1 (pre-infusion and end of infusion), Day 2 (24 hours post Day 1 infusion), Day 8, and Day 15
Population: Participants who were treated with MEDI-575 and for whom serum concentrations were available for PK data analyses. Here "Number of Participants Analyzed" denotes the participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: microgram per milliliter
Groups:
- Carboplatin/Paclitaxel + MEDI-575 - Phase 2: Carboplatin/paclitaxel regimen (carboplatin AUC = 6 mg/mL*min, and paclitaxel 200 mg/m^2) followed by MEDI-575 at a dose of 25 milligram per kilogram (mg/kg) administered as an IV infusion once every 21 days on Day 1 for a total of 6 cycles. Participants who achieved stable disease or better at the completion of carboplatin/paclitaxel therapy and did not demonstrate toxicity to MEDI-575, MEDI-575 alone was continued until unacceptable toxicity, disease progression, initiation of alternative anticancer therapy, or other reasons for participant withdrawal.
Arm/Group | Carboplatin/Paclitaxel + MEDI-575 - Phase 1b | Carboplatin/Paclitaxel + MEDI-575 - Phase 2
Number analyzed (Participants) | 4 | 44
microgram per milliliter | 589.3 (175.6) | 628.9 (441.8)

13. Secondary Outcome: Time of Maximal Observed Concentration (Tmax) of MEDI-575 After First Dose
Description: The tmax refers to the time after dosing when a drug attains its highest measurable concentration (Cmax). The Tmax of MEDI-575 after first dose is reported.
Time Frame: Day 1 (pre-infusion and end of infusion), Day 2 (24 hours post Day 1 infusion), Day 8, and Day 15
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Carboplatin/Paclitaxel + MEDI-575 - Phase 1b | Carboplatin/Paclitaxel + MEDI-575 - Phase 2
Number analyzed (Participants) | 4 | 44
day | 0.044 (0.002) | 0.046 (0.009)

14. Secondary Outcome: Area Under the Concentration-Time Curve Over the Dosing Interval (AUCtau) of MEDI-575 After First Dose
Description: The AUCtau defined as area under the plasma concentration time profile from time zero to the end of the dosing interval (tau). The AUCtau of MEDI-575 after first dose is reported.
Time Frame: Day 1 (pre-infusion and end of infusion), Day 2 (24 hours post Day 1 infusion), Day 8, and Day 15
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: microgram*day per milliliter
Arm/Group | Carboplatin/Paclitaxel + MEDI-575 - Phase 1b | Carboplatin/Paclitaxel + MEDI-575 - Phase 2
Number analyzed (Participants) | 3 | 40
microgram*day per milliliter | 3550 (496.1) | 4803 (1948)

15. Secondary Outcome: Maximum Serum Concentration at Steady State (Cmax,ss) of MEDI-575
Description: The Cmax,ss of MEDI-575 is reported.
Time Frame: Cycle 1 (pre-infusion and end of infusion on Day 1, Day 2, Day 8, and Day 15); Day 1 of Cycles 2 to 4 (pre-infusion and end of infusion)
Population: Participants who were treated with MEDI-575 and for whom serum concentrations were available for PK data analyses. Here "Number of Participants Analyzed" denotes the participants who received at least 4 doses of MEDI-575 and were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: microgram per milliliter
Arm/Group | Carboplatin/Paclitaxel + MEDI-575 - Phase 1b | Carboplatin/Paclitaxel + MEDI-575 - Phase 2
Number analyzed (Participants) | 2 | 27
microgram per milliliter | 2997 (2588) | 619.7 (160.5)

16. Secondary Outcome: Time to Maximum Serum Concentration at Steady State (Tmax,ss) of MEDI-575
Description: The Tmax,ss of MEDI-575 is reported.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Carboplatin/Paclitaxel + MEDI-575 - Phase 1b | Carboplatin/Paclitaxel + MEDI-575 - Phase 2
Number analyzed (Participants) | 2 | 27
day | 0.042 (0.000) | 0.049 (0.017)

17. Secondary Outcome: Trough Serum Concentration at Steady State (Ctrough,ss) of MEDI-575
Description: The Ctrough,ss of MEDI-575 is reported.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: microgram per milliliter
Arm/Group | Carboplatin/Paclitaxel + MEDI-575 - Phase 1b | Carboplatin/Paclitaxel + MEDI-575 - Phase 2
Number analyzed (Participants) | 2 | 28
microgram per milliliter | 375 (155) | 168 (75.6)

18. Secondary Outcome: Percentage of Participants With Positive Anti-MEDI-575 Antibodies
Description: Immunogenicity assessment included determination of anti-drug (MEDI-575) antibodies in serum samples.
Time Frame: Day 1 (prior to infusion) of Cycles 1 to 7 (21-day cycle), end of treatment, 30 and 60 days after the last dose (approximately 3 years)
Population: The evaluable population included all participants who were treated with MEDI-575 and for whom at least one serum sample for immunogenicity testing was available.
Measure: Number; unit: percentage of participants
Arm/Group | Carboplatin/Paclitaxel + MEDI-575 - Phase 1b | Carboplatin/Paclitaxel + MEDI-575 - Phase 2
Number analyzed (Participants) | 4 | 49
percentage of participants | 25.0 (496.1) | 26.5 (1948)

19. Secondary Outcome: Number of Participants With Platelet-derived Growth Factor Receptor Alpha (PDGFRα) Expression in Tumor Cells of Archived Tumor Samples
Description: The immunohistochemical expression of PDGFRα in tumor cells in archived formalin-fixed paraffin-embedded tissue samples collected at baseline are reported. The transmembrane receptor tyrosine kinase PDGFRα plays an important role in human carcinogenesis, both as a direct target on tumor cells and also as a mediator of stromal support for cancer cell growth. The data of positive-staining tumor cells are reported in 3 categories: intensity (1+ [weak expression, staining in <5 % of tumor cells]; 2+ [moderate expression, staining in >= 5 % of tumor cells]; and 3+ [strong expression, staining in >5 % of the tumor cells]), localization (membranous, cytoplasmic, or nuclear), and frequency (rare, occasional, or frequent).
Time Frame: Baseline (Screening [Days -28 to -1])
Population: Evaluable populations for PDGFRα expression included all randomized participants who had formalin-fixed paraffin-embedded samples available at baseline and had positive-staining for tumor cells.
Measure: Count of Participants; unit: Participants
Groups:
- Carboplatin/Paclitaxel - Phase 2: Carboplatin/paclitaxel regimen (carboplatin area under the plasma concentration-time curve [AUC] of 6 milligram per milliliter into minute [mg/mL*min], and paclitaxel 200 milligram per square meter [mg/m^2]) administered as an intravenous (IV) infusion once every 21 days on Day 1, for a total of 6 doses (cycles) or until unacceptable toxicity, disease progression, or other reasons for participant withdrawal.
Arm/Group | Carboplatin/Paclitaxel + MEDI-575 - Phase 1b | Carboplatin/Paclitaxel + MEDI-575 - Phase 2 | Carboplatin/Paclitaxel - Phase 2
Number analyzed (Participants) | 1 | 5 | 3
Participants
  Intensity: 1+ | 1 | 2 | 3
  Intensity: 2+ | 0 | 2 | 0
  Intensity: 3+ | 0 | 1 | 0
  Localization: cytoplasmic | 0 | 3 | 2
  Localization: membranous | 0 | 2 | 0
  Localization: nuclear | 1 | 0 | 1
  Frequency: rare | 1 | 3 | 1
  Frequency: occasional | 0 | 0 | 1
  Frequency: frequent | 0 | 2 | 1

20. Secondary Outcome: Number of Participants With PDGFRα Expression in Stromal Cells of Archived Tumor Samples
Description: The immunohistochemical expression of PDGFRα in stromal cells in archived formalin-fixed paraffin-embedded tissue samples collected at baseline are reported. The transmembrane receptor tyrosine kinase PDGFRα plays an important role in human carcinogenesis, both as a direct target on tumor cells and also as a mediator of stromal support for cancer cell growth. The data of positive-staining stromal cells are reported in 3 categories: intensity (1+ [weak expression, staining in <5 % of tumor cells]; 2+ [moderate expression, staining in >= 5 % of tumor cells]; and 3+ [strong expression, staining in >5 % of the tumor cells]), localization (membranous, cytoplasmic, or nuclear), and frequency (rare, occasional, or frequent).
Time Frame: Baseline (Screening [Days -28 to -1])
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Carboplatin/Paclitaxel + MEDI-575 - Phase 1b | Carboplatin/Paclitaxel + MEDI-575 - Phase 2 | Carboplatin/Paclitaxel - Phase 2
Number analyzed (Participants) | 3 | 16 | 10
Participants
  Intensity: 1+ | 2 | 3 | 3
  Intensity: 2+ | 1 | 10 | 5
  Intensity: 3+ | 0 | 3 | 2
  Localization: cytoplasmic | 3 | 15 | 10
  Localization: membranous | 0 | 1 | 0
  Localization: nuclear | 0 | 0 | 0
  Frequency: rare | 0 | 3 | 1
  Frequency: occasional | 1 | 4 | 3
  Frequency: frequent | 2 | 9 | 6

ADVERSE EVENTS:
Time Frame: From signing of informed consent form until 90 days post the last dose treatment (approximately 3 years)
Arm/Group | Carboplatin/Paclitaxel + MEDI-575 (Total) | Carboplatin/Paclitaxel (Total)
All-Cause Mortality (participants affected / at risk) | 35/53 | 23/43
Serious Adverse Events (participants affected / at risk) | 25/53 | 17/43
Other Adverse Events (participants affected / at risk) | 53/53 | 41/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carboplatin/Paclitaxel + MEDI-575 (Total) (N=53) | Carboplatin/Paclitaxel (Total) (N=43)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (3) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pericolic abscess (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 3 (3)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 4 (5) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (3) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary cavitation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carboplatin/Paclitaxel + MEDI-575 (Total) (N=53) | Carboplatin/Paclitaxel (Total) (N=43)
Anaemia (Blood and lymphatic system disorders) | 24 (73) | 14 (28)
Leukopenia (Blood and lymphatic system disorders) | 6 (23) | 2 (6)
Neutropenia (Blood and lymphatic system disorders) | 12 (37) | 6 (9)
Thrombocytopenia (Blood and lymphatic system disorders) | 10 (46) | 3 (3)
Tachycardia (Cardiac disorders) | 2 (2) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 10 (12) | 2 (2)
Constipation (Gastrointestinal disorders) | 13 (16) | 13 (16)
Diarrhoea (Gastrointestinal disorders) | 24 (49) | 8 (11)
Dyspepsia (Gastrointestinal disorders) | 7 (7) | 4 (4)
Nausea (Gastrointestinal disorders) | 27 (41) | 22 (30)
Stomatitis (Gastrointestinal disorders) | 3 (4) | 3 (5)
Vomiting (Gastrointestinal disorders) | 14 (18) | 8 (11)
Asthenia (General disorders) | 10 (15) | 1 (4)
Fatigue (General disorders) | 31 (54) | 23 (35)
Mucosal inflammation (General disorders) | 4 (4) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2) | 3 (3)
Oedema peripheral (General disorders) | 10 (12) | 0 (0)
Pain (General disorders) | 4 (4) | 3 (3)
Pyrexia (General disorders) | 7 (12) | 4 (4)
Urinary tract infection (Infections and infestations) | 4 (5) | 9 (11)
Fall (Injury, poisoning and procedural complications) | 8 (8) | 1 (1)
Alanine aminotransferase increased (Investigations) | 5 (6) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 4 (9) | 3 (3)
Haemoglobin decreased (Investigations) | 5 (5) | 1 (1)
Neutrophil count decreased (Investigations) | 14 (29) | 5 (6)
Platelet count decreased (Investigations) | 9 (22) | 5 (13)
Weight decreased (Investigations) | 14 (17) | 3 (3)
White blood cell count decreased (Investigations) | 10 (23) | 4 (5)
Decreased appetite (Metabolism and nutrition disorders) | 27 (50) | 11 (22)
Dehydration (Metabolism and nutrition disorders) | 7 (10) | 6 (7)
Hyperglycaemia (Metabolism and nutrition disorders) | 7 (12) | 5 (7)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 7 (9) | 3 (4)
Hypocalcaemia (Metabolism and nutrition disorders) | 6 (9) | 3 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 12 (19) | 8 (9)
Hypomagnesaemia (Metabolism and nutrition disorders) | 20 (42) | 10 (14)
Hyponatraemia (Metabolism and nutrition disorders) | 8 (11) | 4 (4)
Hypophosphataemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 (35) | 13 (22)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (18) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 4 (4)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 17 (33) | 14 (25)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (8) | 6 (6)
Dizziness (Nervous system disorders) | 6 (7) | 3 (4)
Dysgeusia (Nervous system disorders) | 12 (12) | 1 (1)
Headache (Nervous system disorders) | 7 (9) | 4 (4)
Neuropathy peripheral (Nervous system disorders) | 18 (44) | 11 (16)
Paraesthesia (Nervous system disorders) | 5 (6) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 14 (24) | 13 (21)
Anxiety (Psychiatric disorders) | 5 (6) | 2 (2)
Confusional state (Psychiatric disorders) | 6 (10) | 1 (1)
Insomnia (Psychiatric disorders) | 9 (10) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (18) | 6 (6)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 4 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 29 (38) | 21 (27)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (4) | 2 (2)
Hypotension (Vascular disorders) | 7 (7) | 1 (1)

LIMITATIONS AND CAVEATS:
In conjunction with the overall risk-benefit assessment, study was terminated prematurely due to safety concerns.

Change in tumor size outcome measure was not analyzed as per changed planned analysis due to premature termination of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.